CLINICAL TRIAL: NCT04808648
Title: A Single-center, Open-label, Drug-drug Interaction Study of SH-1028 Tablets in Healthy Subjects
Brief Title: The Effect of Itraconazole and Rifampicin on the Pharmacokinetics of SH-1028
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHC013-I-05
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — SH-1028; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole and SH-1028 (Experimental): In the itraconazole study, patients received single-dose SH-1028 200 mg on Days 1 and 12 and itraconazole(200 mg twice daily) on Days 8-14 orally.
  Interventions: Drug: SH-1028; Drug: Itraconazole
- Rifampicin and SH-1028 (Experimental): In the rifampicin study, patients received SH-1028 200mg once daily on Days 1 and 14 and rifampicin 600 mg once daily on Days 8-16
  Interventions: Drug: SH-1028; Drug: Rifampicin

INTERVENTIONS:
Drug: SH-1028 — tablet, oral, 200 mg once daily for day 1 and day 12
Drug: Itraconazole — capsule, oral, 200 mg twice daily for day 8 to day 14
  Arms: Itraconazole and SH-1028
Drug: Rifampicin — capsule, oral, 600 mg once daily for day 8 to day 16
  Arms: Rifampicin and SH-1028

SUMMARY:
This is a phase I study to assess the drug-drug interaction of SH-1028 tablets and Itraconazole/Rifampicin tablets. The study also evaluates the pharmacokinetic and tolerability of SH-1028 tablets in healthy subjects. This study provides evidence for the designing of following clinical trial protocols.

DETAILED DESCRIPTION:
A total of 40 evaluable healthy male subjects will be enrolled in this study.The subjects will be divided into two groups, A and B, with 20 people in each group.

In the itraconazole study (Group A), patients received single-dose SH-1028 200 mg on Days 1 and 12 and itraconazole(200 mg twice daily) on Days 8-14 orally.

In the rifampicin study (Group B), patients received SH-1028 200mg once daily on Days 1 and 14 and rifampicin 600 mg once daily on Days 8-16.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers between the age of 18 to 45 years old (including 18 and 45 years old)
2. Body weight between 50.0 and 80.0 kg, Body mass index between 19.0 and 26.0 kg/m2 (including 19.0 and 26.0 kg/m2);
3. Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant;
4. Promise not to smoke, drink alcohol or drink caffeinated beverages during the trial;
5. Be able to communicate well with the researcher and be able to complete the trial in accordance with the program.
6. Male subjects of reproductive potential with partners will be instructed to,and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 6 months after discontinuing treatment with the investigational product.

Exclusion Criteria:

1. History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder. Or any other disease or physiological condition that may affect the results of the study;
2. Those who have undergone surgery within the first 3 months of the screening period, or who plan to undergo surgery during the study period, or who have previously undergone surgery that may affect drug absorption, distribution, metabolism, and excretion;
3. Subjects with dysphagia or have history of gastrointestinal disorders which affects study drug absorption;
4. Alcohol breath test results greater than 0.0mg/100mL.
5. Urine drug screening (morphine, methamphetamine, ketamine, dimethyldioxyamphetamine, tetrahydrocannabinol) positive;
6. Those who had received the vaccine within 28 days prior to screening, or who planned to receive the vaccine during the trial;
7. Positive test for HBs-Ag, HCV-Ab, HIV-Ab, or syphilis antibody;
8. Allergies, have allergies to drugs or foods; or have known allergies to the components of the investigated drug;
9. Those who smoked daily >5 sticks of cigarette, or the weekly alcohol consumption was higher than 14 units of alcohol (1 unit=10ml or 8g absolute alcohol. 25 ml 40% liquor, 330ml 5% beers, 175ml 12% grape wine are equal to 1.0, 1.5 and 2.0 units of alcohol respectively), or the history of drug abuse and drug abuseor 3 months prior to screening period;
10. Subjects with history of blood donation or massive blood loss (> 200 mL) within 3 months prior to screening;
11. Participated in other clinical trials within 3 months before screening;
12. Use of any drugs that alter liver enzyme activity within 28 days prior to screening;
13. Do not promise not to smoke, not drink alcoholic food or beverages, not consume xanthine-rich foods, not consume grapefruit, dragon fruit, mango, lime, carambola or other products within 24 hours before taking the study drug. Prepared foods or beverages, as well as chocolate, tea, coffee or cola and other special diets that affect the absorption, distribution, metabolism and excretion of drugs;
14. People who have used any medicine (including Chinese herbal medicine and health care products) within two weeks before taking the test drug;
15. History of syncope / needle syncope and intolerable intravenous indwelling needle;
16. Those who have special requirements for diet and cannot follow a unified diet;
17. hose who cannot complete this study because of other reasons, or any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-06 (Estimated); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Blood samples collected on Day 1 and Day 12 (arm 1)/Day 14 (arm 2) at pre-dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours post SH-1028 dose
  Pharmacokinetics of SH-1028 by assessment of maximum plasma concentration
AUC(0-last) | Blood samples collected on Day 1 and Day 12 (arm 1)/Day 14 (arm 2) at pre-dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours post SH-1028 dose
  Pharmacokinetics of SH-1028 by assessment of area under the plasma concentration time curve from zero to last assessed timepoint
AUC(0-∞) | Blood samples collected on Day 1 and Day 12 (arm 1)/Day 14 (arm 2) at pre-dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours post SH-1028 dose
  Pharmacokinetics of SH-1028 by assessment of area under the concentration time curve from time 0 to infinity

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 10 days after last dose
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital with Bengbu Medical College, Bengbu, Anhui, China